CLINICAL TRIAL: NCT01596868
Title: A Randomized, Phase II Trial Comparing Induction Chemotherapy Gemcitabine Plus Cisplatin With Docetaxel Plus Cisplatin Followed by Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma in Northwest China
Brief Title: GP VS TP in the Treatment of Advanced Nasopharyngeal Carcinoma in Northwest China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, Director and Professor of Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mshi
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Nasopharyngeal Squamous Cell Carcinoma; Toxicity Due to Radiotherapy
Keywords: Advanced Nasopharyngeal Carcinoma; treatment; Northwest China
MeSH Terms: interventions — Gemcitabine; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine and Cisplatin (Active Comparator): Drug: gemcitabine and cisplatin The GP regimen consists of gemcitabine at a dose of 1,000 mg/m2 by intravenous (i.v.) infusion over 30 min on day 1 and day 8, and cisplatin 80 mg/m2 by i.v. infusion for 4 h on day 1-3, The regime will be repeated every 3 weeks up to a total of 2-3 courses. Concurrent chemoradiotherapy is administrated with 3 cycles of weekly Cisplatin 80 mg/m2 starting on the first day of IMRT..
  Interventions: Drug: gemcitabine and cisplatin
- docetaxel and cisplatin (Active Comparator): Drug: Docetaxel and cisplatin TP regimen consists of docetaxel at a dose of 75 mg/m2/day on day 1, and cisplatin 80 mg/m2 by i.v. infusion for 4 h on day 1-3. The regime will be repeated every 3 weeks up to a total of 2-3 courses. Concurrent chemoradiotherapy is administrated with 3 cycles of weekly Cisplatin 80 mg/m2 starting on the first day of IMRT.
  Interventions: Drug: docetaxel and cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin — Drug: gemcitabine and cisplatin The GP regimen consists of gemcitabine at a dose of 1,000 mg/m2 by intravenous (i.v.) infusion over 30 min on day 1 and day 8, and cisplatin 80 mg/m2 by i.v. infusion for 4 h on day 1-3, The regime will be repeated every 3 weeks up to a total of 2-3 courses. Concurrent chemoradiotherapy is administrated with 3 cycles of weekly Cisplatin 80 mg/m2 starting on the first day of IMRT.
  Other Names: GP
  Arms: Gemcitabine and Cisplatin
Drug: docetaxel and cisplatin — Drug: Docetaxel and cisplatin The TP regimen consists of docetaxel at a dose of 75 mg/m2/day on day 1,and cisplatin 80 mg/m2 by i.v. infusion for 4 h on day 1-3, The regime will be repeated every 3 weeks up to a total of 2-3 courses. Concurrent chemoradiotherapy is administrated with 3 cycles of weekly Cisplatin 80 mg/m2 starting on the first day of IMRT.
  Other Names: TP
  Arms: docetaxel and cisplatin

SUMMARY:
The present study is a randomized, control, phase II study of locally advanced nasopharyngeal carcinoma (NPC) in Northwest China treated with Gemcitabine plus cisplatin regimen (GP) or Docetaxel plus cisplatin regimen (TP) induction chemotherapy followed by concurrent chemoradiotherapy. The population consists of stage III-IVb nasopharyngeal carcinoma (NPC). The effectiveness, side effects and quality of life will be evaluated according to Standard WHO response criteria, NCI-CTC AE V3.0 and EORTC QLQ-C30 and H&N35 questionnaire.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma has an unique geographic distribution, and has different pathological types, natural history, treatment modalities in endemic and non-endemic regions. Nasopharyngeal carcinoma is both radiosensitive and chemosensitive. Chemoradiotherapy is the main therapy choice for the locoregionally advanced nasopharyngeal carcinoma. However,the optimal chemoradiotherapy regimen has not been determined. Many new drugs including docetaxel and gemcitabine have been incorporated in the induction chemotherapy phase of NPC. The investigators designed the present study with induction chemotherapy follow by CCRT for locoregionally advanced NPC in non-endemic Northwest China, comparing induction chemotherapy regime of TP and GP. The primary objectives were overall response rate (ORR), acute toxicity, tolerance; second objective were overall survival (OS), progression free survival (PFS), rate of distant metastases,late adverse events and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven WHO II~III native NPC in northwest region of China;
* 18 Years to 70 Years;
* stages III-IVb according to AJCC stage classification(7th edition), no previous chemotherapy and radiotherapy;
* Performance status: 0-1(ECOG);
* WBC > 4.0X109/L, PLT > 100X109/L, with normal hepatic function(AST, ALT < 2.5 x upper limit of normal, and bilirubin < 1.5 x upper limit of normal), with normal renal function (Creatinine < 1.5 x upper limit of normal);
* Ability to comply with trial requirements.

Exclusion Criteria:

* Evidence of metastases by clinical or radiographic examinations;
* History of malignancy;
* Prior chemotherapy or anticancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region except for radioactive iodine therapy.;
* Patients with uncontrolled intercurrent disease;
* Patients with currently active malignancy;
* Pregnant or lactating women patients of childbearing potential who are unwilling to practice adequate contraception during study treatment and for two months after the last administration of study drug.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
overall response rate (ORR) | 3-year

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Locoregional failure-free survival | 3-year
  the date of randomization to the first local failure
Distant failure-free survival | 3-year
  from randomization to the first remote failure
Number of Participants with Adverse Events | 3-year
Quality of life | 3-year
Acute adverse reaction | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Mei Shi, MD, Principal Investigator — department of radiation oncology
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military, Xi’an, Shanxi, China